CLINICAL TRIAL: NCT00180167
Title: Therapy of AML in Patients Older Than 60 Years: Randomized Comparison of a Double Induction With Daunorubicin and AraC (as Continuous Infusion) With a Double Induction With Mitoxantrone and Intermittent, Medium High Dose AraC
Brief Title: Therapy of Acute Myeloid Leukemia in Patients Over the Age of 60 : DA Versus Mitoxantrone With Intermittent AraC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Technische Universität Dresden (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AML_GT60_DD
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2010-08-20 (Estimated); Status verified 2010-08

CONDITIONS: Leukemia, Nonlymphocytic, Acute
Keywords: Chemotherapy; elderly
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Daunorubicin + Ara-C (Active Comparator)
  Interventions: Drug: randomization between two established Chemotherapies
- Mitoxantrone + Ara-C (Experimental)
  Interventions: Drug: randomization between two established Chemotherapies

INTERVENTIONS:
Drug: randomization between two established Chemotherapies

SUMMARY:
Single Arm-Studies suggest improved remission and survival rates for a Protocol with Mitoxantron 10mg/m2 for 3 days combined with AraC 1g/m2 bid on days 1+3+5+7 compared to a conventional DA 7+3 protocol (45mg/m2 Daunorubicin).

DETAILED DESCRIPTION:
Randomized comparison of the two protocols.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of AML
* age >60
* no previous Chemo for AML
* informed consent
* Karnofsky >70

Exclusion Criteria:

* AML M3
* uncontrolled Sepsis
* uncontrolled HYpertension
* respiratory failure
* heart-failure NYHA IV, recent myocardial infarction
* severe organ dysfunction of liver, kidneys,
* HIV -infection or active Hepatitis B,C

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 492 (Actual)
Dates: Start 2005-01; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Complete remission rate
Survival

SECONDARY OUTCOMES:
toxicity
Secondary purpose: Is the prognostic evaluation of the treating physician prior to initiation of chemotherapy (prior to randomization) of predictive value?

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich S. Schuler, PD Dr. med., Principal Investigator — University Hospital Dresden, Germany
Locations (1):
- Universitätsklinikum, Dresden, Saxony, Germany

REFERENCES:
- [Background] Mantovani L, Hasenclever D, Krahl R, Ponisch W, Herold M, Pasold R, Fiedler F, Dolken G, Kampfe D, Schmoll HJ, Subert R, Kubel M, Niederwieser D, Helbig W; East German Hematology and Oncology Group (OSHO). Intermediate-dose cytarabine treatment delivered at moderate infusion rates for de novo acute myeloid leukemia-results of a phase I-II study. Leuk Lymphoma. 2002 Feb;43(2):265-74. doi: 10.1080/10428190290006035. PMID 11999557
- [Derived] Kunadt D, Stasik S, Metzeler KH, Rollig C, Schliemann C, Greif PA, Spiekermann K, Rothenberg-Thurley M, Krug U, Braess J, Kramer A, Hochhaus A, Scholl S, Hilgendorf I, Brummendorf TH, Jost E, Steffen B, Bug G, Einsele H, Gorlich D, Sauerland C, Schafer-Eckart K, Krause SW, Hanel M, Hanoun M, Kaufmann M, Wormann B, Kramer M, Sockel K, Egger-Heidrich K, Herold T, Ehninger G, Burchert A, Platzbecker U, Berdel WE, Muller-Tidow C, Hiddemann W, Serve H, Stelljes M, Baldus CD, Neubauer A, Schetelig J, Thiede C, Bornhauser M, Middeke JM, Stolzel F; A. M. L. Cooperative Group (AMLCG), Study Alliance Leukemia (SAL). Impact of IDH1 and IDH2 mutational subgroups in AML patients after allogeneic stem cell transplantation. J Hematol Oncol. 2022 Sep 5;15(1):126. doi: 10.1186/s13045-022-01339-8. PMID 36064577